CLINICAL TRIAL: NCT00488982
Title: A Randomized Phase II Study of Intermittent Chemotherapy or Intermittent Chemotherapy With Maintenance GM-CSF in Patients With Previously Untreated Hormone Refractory Prostate Cancer
Brief Title: Intermittent Chemotherapy With or Without Granulocyte-macrophage Colony-stimulating Factor (GM-CSF) for Metastatic Hormone Refractory Prostate Cancer (HRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 055511; NCI-2011-01269 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: Metastatic Hormone Refractory Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Docetaxel + Observation (Experimental): Intermittent docetaxel/prednisone with no maintenance therapy: Patients will discontinue docetaxel/prednisone and undergo observation until disease progression at which time they will re-initiate docetaxel/prednisone. Six cycles of docetaxel/prednisone will again be administered before subsequent discontinuation of chemotherapy
  Interventions: Drug: Docetaxel
- Docetaxel + GM-CSF (Experimental): Intermittent docetaxel/prednisone with maintenance GM-CSF therapy: Patients will discontinue docetaxel/prednisone and will receive maintenance GM-CSF until disease progression at which time, they will discontinue GM-CSF and resume docetaxel/prednisone. Six cycles of docetaxel/prednisone will again be administered before discontinuation of chemotherapy and GM-CSF therapy is re-initiated. GM-CSF dose/schedule will be as previously described (250 mcg/m2 SQ daily, days 15-28 q28 days)
  Interventions: Drug: Docetaxel and GM-CSF

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75mg/m2 every 21 days
  Arms: Docetaxel + Observation
Drug: Docetaxel and GM-CSF — Docetaxel 75mg/m2 every 21 days and GM-CSF 250mcg/m2 SQ days 15-28
  Arms: Docetaxel + GM-CSF

SUMMARY:
This is a two-arm, randomized Phase II study of intermittent chemotherapy with and without GM-CSF. All patients will receive six 21-day cycles of docetaxel 75 mg/m2 on Day 2 of each cycle and 5 mg prednisone twice a day on Days 1-21. Following six cycles of chemotherapy, eligible subjects will be randomized to no maintenance therapy or to maintenance GM-CSF therapy. The GM-CSF group dose schedule will be 250 mcg/m2 subcutaneous (SQ) daily Days 15-28 every 28 days. Patients in both groups will continue until disease progression at which time GM-CSF will be discontinued and chemotherapy will again be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years
2. Histologically documented adenocarcinoma of the prostate
3. Progressive metastatic prostate cancer
4. Castrate levels of testosterone (<50 ng/ml) must be maintained
5. Prior hormonal therapy or medications :

   Patients who are receiving an anti-androgen, secondary hormonal therapy (i.e. ketoconazole, aminoglutethimide, megestrol acetate, diethylstilbestrol), 5-alpha reductase inhibitor (i.e. finasteride (Proscar), dutasteride (Avodart)) or herbal prostate medication (i.e. saw palmetto, PC-SPES, PC-PLUS) must discontinue the drug by the date of initiation of chemotherapy on study
6. ≥ 4 weeks since major surgery and fully recovered
7. ≥ 4 weeks since any prior radiation with any toxicity attributable to radiation resolved to ≤grade 1
8. ≥ 8 weeks since the last dose of strontium or samarium
9. Sexually active patients must agree to use adequate contraception
10. Karnofsky Performance Status ≥ 60%
11. Life expectancy >12 weeks
12. Required initial laboratory values Absolute neutrophil count > 1500/ul Platelets > 100,000/ul Hemoglobin > 8.0 g/dl Creatinine ≤ 2.0 X upper limit of normal Bilirubin ≤upper limit of normal (ULN)

aspartate aminotransferase (AST) / alanine aminotransferase (ALT) / alkaline phosphatase: AST AND ALT AND alkaline phosphatase must be within the range allowing for eligibility In determining eligibility, the more abnormal of the 2 values (AST or ALT should be used. An abnormal alkaline phosphatase must be attributed to liver dysfunction and not metastatic bone involvement (i.e elevated gamma-glutamyl transpeptidase (GGTP) or evidence of liver metastases)

Inclusion criteria for late enrolling patients:

1. Age over 18 years
2. Histologically documented adenocarcinoma of the prostate
3. ≤3 cycles of prior docetaxel chemotherapy for metastatic disease permitted prior to enrollment
4. Docetaxel must have been administered on an every 3 week schedule
5. Each docetaxel dose must have been between 60 and 75 mg/m2
6. Castrate levels of testosterone <50 ng/mL
7. Daily use of other steroids (hydrocortisone, dexamethasone) instead of prednisone or no steroids, is permitted up until time of enrollment
8. A Prostate-specific antigen (PSA) level must have been documented within 6 weeks of initiating docetaxel chemotherapy

Exclusion Criteria:

1. Prior systemic chemotherapy for prostate cancer, other than q 3-week docetaxel/prednisone. Prior neoadjuvant or adjuvant chemotherapy is permitted if there was no evidence of disease relapse within 12 months of the last dose of chemotherapy.
2. >3 cycles of q3 week docetaxel/prednisone chemotherapy has already been administered to the patient
3. Peripheral neuropathy >grade 1
4. Prior immunotherapy including systemic GM-CSF or vaccines utilizing GM-CSF; prior G-CSF support of chemotherapy-related neutropenia is permitted
5. Prior biologic agents (i.e.,anti-angiogenic agents, anti-Epithelial Growth Factor Receptor (EGFR) inhibitors)≤ 4 weeks prior to registration
6. More than two prior therapies with an investigational agent, completed ≤ 4 weeks prior to enrollment (no prior immunotherapeutics are allowed)
7. Myocardial infarction or significant change in anginal pattern within the last 6 months, symptomatic congestive heart failure (NYHA Class III or higher) or uncontrolled cardiac arrhythmia
8. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded
9. Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 will be excluded
10. Poorly controlled diabetes (fasting blood glucose >250) despite optimization of medical therapy

Exclusion criteria for late enrolling patients:

1. Prior immunotherapy including systemic GM-CSF or vaccines utilizing GM-CSF; prior G-CSF support for chemotherapy-related neutropenia is permitted
2. Delay of ≥6 weeks between any 2 chemotherapy cycles prior to enrollment on study
3. Cumulative delays ≥8 weeks between chemotherapy cycles prior to enrollment on study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-04; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Small, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - University of California, San Francisco, San Francisco, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health and Science University Cancer Institute, Portland, Oregon
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients had to complete 6 cycles of induction chemotherapy and have a ≥ 50% decline in prostate-specific antigen to be eligible for randomization.
Groups:
- Pre-Randomization: Induction chemotherapy for 6 cycles (1 cycle = 21 days)
  * Docetaxel 75mg/m^2 I.V. (intravenous) on day 2
  * Prednisone 5 mg by mouth (p.o.), twice a day (b.i.d.) from day 1 to 21 (for 21 days)
- Docetaxel and Observation: Docetaxel 75mg/m^2 every 21 days
- Docetaxel and GM-CSF: Docetaxel 75mg/m^2 every 21 days and GM-CSF 250mcg/m^2 subcutaneously days 15-28
Period: Induction Chemotherapy
Arm/Group | Pre-Randomization | Docetaxel and Observation | Docetaxel and GM-CSF
Started | 125 | 0 | 0
6 Cycles Completed | 94 | 0 | 0
≥ 50% Prostate-specific Antigen Decline | 52 | 0 | 0
Completed | 52 | 0 | 0
Not Completed | 73 | 0 | 0
Period: Course 1
Arm/Group | Pre-Randomization | Docetaxel and Observation | Docetaxel and GM-CSF
Started | 0 | 25 | 27
Completed | 0 | 13 | 13
Not Completed | 0 | 12 | 14
Not completed — Physician Decision | 0 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 8 | 2
Not completed — nonprotocol therapy | 0 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 6
Period: Course 2
Arm/Group | Pre-Randomization | Docetaxel and Observation | Docetaxel and GM-CSF
Started | 0 | 13 | 13
Completed | 0 | 4 | 8
Not Completed | 0 | 9 | 5
Period: Course 3
Arm/Group | Pre-Randomization | Docetaxel and Observation | Docetaxel and GM-CSF
Started | 0 | 4 | 8
Completed | 0 | 2 | 3
Not Completed | 0 | 2 | 5
Period: Response to Course 3
Arm/Group | Pre-Randomization | Docetaxel and Observation | Docetaxel and GM-CSF
Started | 0 | 2 | 3
Completed | 0 | 1 | 0
Not Completed | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: * Induction Chemotherapy: Total number of patients enrolled, starting trial.
  * Docetaxel/Docetaxel and GM-CSF: patients which passed 6 cycles of induction chemotherapy and had a ≥ 50 % PSA decline
Groups:
- All Patients Accrued: There were a total of 125 patients whom were accrued to the study and assigned to at least one course of docetaxel
Arm/Group | All Patients Accrued
Number analyzed (Participants) | 125
Age, Customized [Median (Full Range); unit: years]
  Median Age Range | 70 [47 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 125
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 115
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 111
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 125
Gleason Score [Count of Participants; unit: Participants] — The Gleason Score ranges from 1-8. Scores of 1-5 describe how much the cancer from a biopsy looks like healthy tissue (lower score) or abnormal tissue (higher score). Typical Gleason Scores range from 6-10. The higher the Gleason Score, the more likely that the cancer will grow and spread quickly. Since prostate tumors are often made up of cancerous cells with different grades, two grades are assigned for each patient. A primary grade for cells that make up the largest area of tumor and a secondary grade for cells of next largest area. Together they make up the total Gleason Score.
  Participants
    <=6 | 22
    7 | 33
    8-10 | 70

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: The Kaplan-Meier product limit method with 95% confidence intervals will be used to estimate the median time to disease progression during initial course of randomized treatment
Time Frame: Up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Docetaxel and Observation: - Docetaxel 75mg/m^2 every 21 days
- Docetaxel and GM-CSF: * Docetaxel 75mg/m^2 every 21 days
  * GM-CSF 250mcg/m2 subcutaneous (SQ) days 15-28
Arm/Group | Docetaxel and Observation | Docetaxel and GM-CSF
Number analyzed (Participants) | 25 | 27
months | 1.5 [1.5 to 2.4] | 3.3 [2.4 to 3.5]

2. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier product limit method will be used to estimate the median overall survival
Time Frame: Up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Docetaxel and Observation: Docetaxel 75mg/m2 every 21 days
- Docetaxel and GM-CSF: Docetaxel 75mg/m2 every 21 days GM-CSF 250mcg/m2 SQ days 15-28
- Overall Survival: Includes all patients whom received any treatment starting with first course of Docetaxel at Induction
Arm/Group | Docetaxel and Observation | Docetaxel and GM-CSF | Overall Survival
Number analyzed (Participants) | 25 | 27 | 125
months | 14 [10.5 to 27.6] | 28.4 [19.2 to 34.1] | 15.6 [13.1 to 18.8]

3. Secondary Outcome: Number of Participants With PSA Response to Successive Series of Chemotherapy
Description: PSA partial response is defined by at least a 50% decline from PSA value from the baseline measurement to 12 weeks of protocol therapy. The decline must be confirmed by a second PSA value obtained 4 or more weeks later For those patients whose PSA have decreased but has not reached response criteria defined above, progressive disease is defined as 25% increase over the nadir PSA value provided that the increase is at least 5ng/mL and is confirmed.
Time Frame: Up to 6 years
Population: Twenty-six participants total resumed a second course of the Docetaxel, and five participants went on to resume a third course of treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Docetaxel and Observation: - Docetaxel 75mg/m2 every 21 days
- Docetaxel and GM-CSF: * Docetaxel 75mg/m2 every 21 days
  * GM-CSF 250mcg/m2 SQ days 15-28
Arm/Group | Docetaxel and Observation | Docetaxel and GM-CSF
Number analyzed (Participants) | 13 | 13
Participants
  PSA response to Course 2 chemotherapy | 4 | 8
  PSA response to Course 3 chemotherapy: number analyzed (Participants) | 2 | 3
  PSA response to Course 3 chemotherapy | 1 | 0

4. Secondary Outcome: Cumulative Duration of Time on and Off Docetaxel-based Therapy
Description: Median percentage of time will be calculated to summarize the total duration of chemotherapy and amount of docetaxel/prednisone administered while the patient is on study. The same results will be tabulated for each. For the on-chemotherapy period: will be estimated from the date of starting protocol therapy; if a patient received docetaxel on day 2 of a cycle, he will be considered to have received a full 21 days on therapy. For the off-chemotherapy period: will be calculated from the date of starting the observation or GM-CSF period to the date of resuming chemotherapy
Time Frame: Up to 7 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Docetaxel and Observation OFF Chemotherapy: Starting the docetaxel with observation period to date of resuming chemotherapy post initial induction
- Docetaxel and GM-CSF OFF Chemotherapy: Starting the docetaxel with GM-CSF period to date of resuming chemotherapy post initial induction
- Docetaxel + Observation ON Chemotherapy: Starting Docetaxel 75mg/m2 and Observation every 21 days for at least 2 days
- Docetaxel and GM-CSF ON Chemotherapy: Starting Docetaxel 75mg/m2 and GM-CSF 250mcg/m2 SQ days 15-28 every 28 days with at least 2 days of Docetaxel
Arm/Group | Docetaxel and Observation OFF Chemotherapy | Docetaxel and GM-CSF OFF Chemotherapy | Docetaxel + Observation ON Chemotherapy | Docetaxel and GM-CSF ON Chemotherapy
Number analyzed (Participants) | 25 | 27 | 25 | 27
months | 24.7 [0.8 to 50.8] | 30.9 [1.7 to 77.1] | 8.3 [3.9 to 22.8] | 7.6 [1.9 to 19.2]

ADVERSE EVENTS:
Time Frame: Any patient receiving at least one dose of the study treatment will be included in the analyses of toxicity during the initial chemotherapy period, but patients who cancel registration before receiving any therapy will not. All grade 3-5, expected and unexpected adverse events (AEs) were collected at all study visits from time of first treatment until at least 28 days following the last dose of study drug.
Description: Data was not collected per intervention. All patients were assigned to the same treatment of Docetaxel/Prednisone before being assigned to the subsequent therapy arms where they may have received multiple treatment courses with multiple inductions. Abnormal lab values or test results constituted AEs only if they induced clinical signs /symptoms, required therapy, or required dose modification. There were no treatment-associated deaths.
Groups:
- All Accrued Patients: All patients were assigned to received six 21-day cycles of docetaxel 75 mg/m2 on Day 2 of each cycle and 5 mg prednisone twice a day on Days 1-21. Following six cycles of chemotherapy, eligible subjects were randomized to no maintenance therapy or to maintenance GM-CSF therapy. Patients in both groups were followed until disease progression at which time GM-CSF was discontinued and another course of docetaxel and prednisone was administered again.
Arm/Group | All Accrued Patients
All-Cause Mortality (participants affected / at risk) | 8/125
Serious Adverse Events (participants affected / at risk) | 20/125
Other Adverse Events (participants affected / at risk) | 0/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Accrued Patients (N=125)
Febrile neutropenia (Infections and infestations) | 8 (9)
Neutropenia (Infections and infestations) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes